CLINICAL TRIAL: NCT02819440
Title: PDE5 Inhibition for Obesity-Related Cardiometabolic Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Evan Brittain, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 160208
Record Dates: First submitted 2016-06-21; First posted 2016-06-30 (Estimated); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Healthy; Obese
MeSH Terms: conditions — Obesity | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Active Comparator): Subjects will be randomized to one of two arms. 100 obese adult subjects will be randomized to the Tadalafil arm following the screening visit. Beginning at their baseline visit, they will receive an oral daily dose of Tadalafil (20mg) that they will take for 12 weeks (through their completion of the study). After randomization has occurred, the active comparator subjects will undergo the following visit protocol: baseline visit (two half-days), an interim visit (6 weeks post-baseline), and a 12-week visit (two half-days).
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Subjects will be randomized to one of two arms. 100 obese adult subjects will be randomized to the placebo arm following the screening visit. Beginning at their baseline visit, they will receive an oral daily dose of a placebo pill (20mg) that they will take for 12 weeks (through their completion of the study). After randomization has occurred, the placebo comparator subjects will undergo the following visit protocol: baseline visit (two half-days), an interim visit (6 weeks post-baseline), and a 12-week visit (two half-days).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — Tadalafil is an FDA approved, clinically-available drug that inhibits the enzyme phosphodiesterase type 5A (PDE5). Subjects who are randomized to this arm will be provided with 20mg of Tadalafil to take every day for 12 weeks, beginning at their baseline visit.
  Other Names: CIALIS
  Arms: Tadalafil
Drug: Placebo — 100 patients will be randomized to receive a placebo pill. Subjects in this arm will be provided with 20mg Placebo to take every day for 12 weeks, beginning at their baseline visit.
  Arms: Placebo

SUMMARY:
Obesity and its adverse cardiometabolic consequences are major public health problems. Several features of obesity contribute to the associated cardiovascular risk and are potential targets for intervention. These include insulin resistance and beta cell dysfunction, reduced metabolic rate, and impaired aerobic capacity.The purpose of this study is to examine if the phosphodiesterase type 5A inhibitor tadalafil improves cardiometabolic health in individuals who are obese and insulin resistant.

DETAILED DESCRIPTION:
Obesity is a risk factor for nearly all cardiovascular (CV) disease including coronary artery disease, hypertension, and heart failure. Increased CV risk in obese individuals appears to depend largely on the degree of metabolic dysregulation and metabolic risk factors (glucose intolerance, dyslipidemia, etc.). Notably, interventions that improve insulin sensitivity and cardiorespiratory fitness can reduce CV risk in obese individuals, even in the absence of weight loss.

The cyclic guanylate monophosphate pathway (cGMP) is involved in energy homeostasis and systemic metabolism. Multiple lines of evidence suggest that increasing cGMP activity is beneficial from a metabolic standpoint. Tadalafil is a clinically-available drug that inhibits the enzyme that breaks down cGMP.

The study investigators hypothesize that chronic PDE5 inhibition in obese, insulin-resistant adults will improve cardiometabolic health.

Aim 1: To examine the effect of PDE5 inhibition on energy expenditure. Aim 2: To examine the effect of PDE5 inhibition on insulin sensitivity and secretion.

Aim 3: To examine the effect of PDE5 inhibition on cGMP tone and circulating mediators of cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 21-50)
* Obesity (BMI ≥ 30 kg/m2)
* Prediabetes on oral glucose tolerance test.

Exclusion Criteria:

* Age <21 or > 50
* BMI < 30 kg/m2
* Systolic blood pressure (SBP) < 100, > 150 mmHg
* Current anti-hypertensive medication use, including diuretics
* Current use of organic nitrates
* Current use of PDE-5 inhibitors (sildenafil, tadalafil, vardenafil)
* History of reaction to PDE-5 inhibitors
* Known HIV infection
* Use of medications that strongly alter CYP3A4 activity
* History of myocardial infarction, angina, uncontrolled cardiac arrhythmia, stroke, transient ischemic attack, or seizure
* Known non-arteritic ischemic optic retinopathy (NAIOR)
* History of hearing loss
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2 by the modified diet in renal disease (MDRD) equation
* Hepatic transaminase (AST and ALT) levels greater than three times the upper limit of normal
* Known pregnancy or breastfeeding or those unwilling to avoid pregnancy during the course of the study
* History of priapism
* Use in excess of four alcoholic drinks daily
* History of diabetes mellitus or use of anti-diabetic medications
* Known anemia (men, Hct < 38% and women, Hct <36%)
* Menopause
* Inability to exercise on a bicycle
* Weight > 300 pounds

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2016-07; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan L Brittain, MD, MSCI, Principal Investigator — Vanderbilt Cardiovascular Medicine; Thomas J Wang, MD, Principal Investigator — Vanderbilt Cardiovascular Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 141 participants passed our screening procedures and were enrolled however only 125 were randomized due to dropouts and scheduling conflicts. We allowed up to 30 days between the screening process and the baseline visit. Participants were assigned to a group after the baseline visit.
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 61 | 64
Completed | 48 | 52
Not Completed | 13 | 12
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 61 | 64 | 125
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.5 (7.8) | 36.0 (8.2) | 36.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 87
  Male | 18 | 20 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 58 | 57 | 115
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 12 | 16 | 28
  White | 46 | 42 | 88
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 64 | 125

OUTCOME MEASURES:

1. Primary Outcome: Resting Energy Expenditure After 12 Weeks of Drug Therapy (kcal/Day)
Description: Subjects will undergo a metabolic chamber protocol to measure resting exercise energy expenditure (kcal/min) at 12 weeks adjusted statistically for the baseline measurement.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 48 | 52
kcal/day | 1267 (133) | 1268 (164)

2. Primary Outcome: Insulin Sensitivity After 12 Weeks of Drug Therapy
Description: Subjects will undergo an insulin modified fasting intravenous glucose tolerance test (FS-IVGTT) protocol at 12 weeks adjusted statistically for the baseline measurement.
Time Frame: 12 weeks
Population: Missing data from 2 participants in the Tadalafil arm, 5 participants in the placebo arm caused by inability to obtain intravenous access, which is necessary to make measurements for this endpoint.
Measure: Median (Inter-Quartile Range); unit: ml/kg/min/μIU ml
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 46 | 47
ml/kg/min/μIU ml | 1.4 [1.0 to 2.3] | 1.5 [0.9 to 1.9]

3. Secondary Outcome: Physical Activity-induced Energy Expenditure (kcal/Day)
Description: During the metabolic chamber protocol, conducted at baseline and at 12 weeks, the cardiopulmonary exercise test protocol will be conducted. The Energy Expenditure (EE) related to physical activity will be calculated as peak EE above the resting level while performing the exercise test.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 48 | 52
kcal/day | 3320 (866) | 3269 (714)

4. Secondary Outcome: Dual Energy X-Ray Absorptiometry (DEXA) (g)
Description: fat mass at 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 48 | 52
grams | 47 (12) | 50 (12)

5. Secondary Outcome: Quality of Life Using the Medical Outcomes Study Short-Form Health Survey (SF-36) Physical Component Score
Description: Quality of life will be assessed using the Medical Outcomes Study Short-Form Health Survey (SF-36). The SF-36 is a 36 question survey with a total score range from 0-100; higher scores indicate better quality of life.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 48 | 52
score on a scale | 52.7 (5.6) | 51.0 (6.9)

6. Secondary Outcome: Change in cGMP/NP Ratio After 12 Weeks of Drug Therapy
Description: Subjects will undergo a fasting blood draw at baseline and 12 weeks to measure the change in ratio of plasma cyclic guanylate monophosphate pathway (cGMP) to plasma natriuretic peptides (NP) in response to the drug intervention (placebo or tadalafil).
Time Frame: 12 weeks
Population: Due to lack of funding, the assays required to measure the participant samples were not performed and there is no data to report.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Maximal Oxygen Consumption
Description: Subjects will undergo a symptom-limited cardiopulmonary exercise test to measure peak oxygen consumption (VO2 max). Maximal oxygen consumption will be measured as 'mL/min'.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 48 | 52
mL/min | 883 (142) | 893 (186)

8. Secondary Outcome: Sexual Function
Description: The Female Sexual Function Index will be used to measure sexual function in women with a range from 2-36 with higher scores indicating better sexual function.
Time Frame: 12 weeks
Population: Test only performed in women as designed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 28 | 35
score on a scale | 23.9 (6.9) | 19.8 (8.9)

9. Secondary Outcome: Maximal Exercise Energy Expenditure (kcal/Day)
Description: Subjects will undergo a metabolic chamber protocol to measure maximal exercise energy expenditure (kcal/min) at 12 weeks adjusted statistically for the baseline measurement. Maximal Exercise Energy Expenditure will be measured as "kcal/day"
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 48 | 52
kcal/day | 4535 (760) | 4588 (976)

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Tadalafil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/64
Other Adverse Events (participants affected / at risk) | 36/61 | 19/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tadalafil (N=61) | Placebo (N=64)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Blood in stool (Gastrointestinal disorders) | 0 | 1
Vaginal spotting/breakthrough bleeding (Reproductive system and breast disorders) | 1 | 1
Elevated liver enzymes (Hepatobiliary disorders) | 0 | 1
Extremity pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Facial cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
Flu (Infections and infestations) | 0 | 1
Fluid retention (Renal and urinary disorders) | 2 | 0
Hair loss (Skin and subcutaneous tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 5
Heartburn (Gastrointestinal disorders) | 5 | 0
Erections (Reproductive system and breast disorders) | 1 | 0
Foot pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 4 | 0
Arm tingling (Musculoskeletal and connective tissue disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Nosebleed (Blood and lymphatic system disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Thrush (Gastrointestinal disorders) | 0 | 1
Tonsilitis (Gastrointestinal disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT02819440/Prot_SAP_000.pdf